CLINICAL TRIAL: NCT05220410
Title: The Safety and Efficacy of Psilocybin in Patients With Treatment-resistant Depression and Chronic Suicidal Ideation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: COMPASS Pathways (Industry)
Responsible Party: Principal Investigator, Scott T. Aaronson, M.D, Director, Clinical Research Programs, Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49348
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-07

CONDITIONS: Treatment Resistant Depression; Suicidal Ideation
Keywords: Psilocybin; Psychedelic; Major depression; Treatment resistant depression; Suicidal ideation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Suicidal Ideation; Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 25mg of Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Open-Label

SUMMARY:
This study aims to explore the safety and tolerability of a single dose of psilocybin (25mg) administered under supportive conditions to adult participants with TRD and chronic suicidal ideation

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age at Screening
* Diagnosis of Major Depressive Disorder (MDD)
* Significant level of suicidal thoughts with active ideation and without immediate intent
* Failure to respond to 2 medications in the current episode

Exclusion Criteria:

* Current or past history of schizophrenia, psychotic disorder, bipolar disorder, borderline personality disorder, etc.
* Current alcohol or substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Modified Scale for Suicidal Ideation (MSSI) | Baseline (V2) to Day 1 (V4), Week 1 (V5), Week 2 (V6), Week 3 (V7), Week 6 (V8), Week 9 (V9) and Week 12 (V10)
  The MSSI is an 18-item clinician rated scale to assess the presence or absence of suicide ideation and the degree of severity of suicidal ideas. Each of the 18 items is rated on a scale of 0 to 3 where a higher score indicates greater suicidal severity.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Baseline (V2) to Day 1 (V4), Week 1 (V5), Week 2 (V6), Week 3 (V7), Week 6 (V8), Week 9 (V9), and Week 12 (V10)
  The MADRS is a clinician rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity.
Concise Health Risk Tracking Self Report 12 Items (CHRT-SR) | Baseline (V2) to Day 1 (V4), Week 1 (V5), Week 2 (V6), Week 3 (V7), Week 6 (V8), Week 9 (V9) and Week 12 (V10)
  The CHRT-SR is a 12-item self-report measure that systematically assesses both suicidal thinking and associated thoughts that might indicate the propensity for suicidal acts.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (V2) to Day 1 (V4), Week 1 (V5), Week 2 (V6), Week 3 (V7), and Week 12 (V10)
  The C-SSRS is a semi-structured interview designed to assess the severity and intensity of suicidal ideation, suicidal behavior, and non-suicidal self injurious behavior over a specified time period. The measurement of suicidal ideation is based on five "yes" or "no" questions with accompanying descriptions arranged in order of increasing severity.
Clinical Global Impression - Modified for Depression (CGI-D) | Baseline (V2) to Week 3 (V7) and Week 12 (V10)
  The CGI is a 3-item observer-rated scale that measures illness severity, global improvement or change and therapeutic response.
Clinical Global Impressions - Modified for Suicidal Ideation (CGI-SI) | Baseline (V2) to Week 3 (V7), and Week 12 (V10)
  The CGI is a 3-item observer-rated scale that measures illness severity, global improvement or change and therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Aaronson, MD, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No